CLINICAL TRIAL: NCT03664557
Title: Feasibility of Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in Patients Suffering From Refractory Cardiac Arrest: a Pilot Study
Brief Title: Feasibility of REBOA in Refractory Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ReaReboa
Record Dates: First submitted 2018-08-31; First posted 2018-09-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Heart Arrest
Keywords: Resuscitation; REBOA
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Open label feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ER Reboa TM Catheter (Experimental): During cardiac arrest occlusion of descending aorta to redistribute CPR-generated blood flow to brain and coronaries
  Interventions: Device: ER Reboa TM Catheter

INTERVENTIONS:
Device: ER Reboa TM Catheter — During cardiac arrest occlusion of descending aorta to redistribute CPR-generated blood flow to brain and coronaries

SUMMARY:
Outcome after non-traumatic cardiac arrest remains poor despite many efforts in improving immediate advanced life support (ALS) and post-arrest therapy. Preserving myocardial and cerebral perfusion in the event of cardiac arrest by the means of effective cardio-pulmonary resuscitation (CPR) is of utmost importance. During CPR, coronary perfusion pressure is a significant predictor of increased rates of return of spontaneous circulation (ROSC) and survival to hospital discharge, while cerebral perfusion pressure is crucial for good neurologic outcome. The absence of ROSC despite prolonged high quality and efficient initial basic life support (BLS) followed by traditional ALS ends finally in neuronal damage and death. Occlusion of the aorta using a REBOA catheter in the management of noncompressible abdominal or pelvic hemorrhage has shown improvements in hemodynamic profiles and has proved to be feasible in both, clinical and preclinical settings for trauma patients in hemorrhagic shock. Animal models of continuous balloon occlusion of the aorta in non-traumatic cardiac arrest have shown meaningful increases in coronary artery blood flow, coronary artery perfusion pressure and carotid blood flow, leading to improved rates of ROSC, 48h-survival and neurological function. These promising data provide an opportunity to improve outcome after cardiac arrest in humans too. Before testing such an approach in humans, the safe and reliable placement procedure of the catheter-balloon in humans after cardiac arrest needs to be established under ongoing CPR.

DETAILED DESCRIPTION:
Background and Rationale Outcome after non-traumatic cardiac arrest remains poor despite many efforts in improving immediate advanced life support (ALS) and post-arrest therapy. Preserving myocardial and cerebral perfusion in the event of cardiac arrest by the means of effective cardio-pulmonary resuscitation (CPR) is of utmost importance. During CPR, coronary perfusion pressure is a significant predictor of increased rates of return of spontaneous circulation (ROSC) and survival to hospital discharge, while cerebral perfusion pressure is crucial for good neurologic outcome. The absence of ROSC despite prolonged high quality and efficient initial basic life support (BLS) followed by traditional ALS ends finally in neuronal damage and death. Occlusion of the aorta using a REBOA catheter in the management of non-compressible abdominal or pelvic haemorrhage has shown improvements in hemodynamic profiles and has proved to be feasible in a preclinical setting for trauma patients in haemorrhagic shock. Animal models of continuous balloon occlusion of the aorta in non-traumatic cardiac arrest have shown meaningful increases in coronary artery blood flow, coronary artery perfusion pressure and carotid blood flow leading to improved rates of ROSC, 48h-survival and neurological function. These promising data provide an opportunity to improve outcome after cardiac arrest in humans too. Before testing such an approach in humans, the safe and reliable placement procedure of the catheter-balloon in humans after cardiac arrest needs to be established under ongoing CPR.

Investigational Product (treatment, device) and Indication The ER-REBOA™ Catheter, Prytime Medical, 229 North Main Street, Boerne, TX 78006, USA, has a CE Declaration of Conformity and is intended, as defined in the instruction manual, for temporary occlusion of large vessels and blood pressure monitoring. The ER-REBOA™ Catheter is specifically designed for use in the emergency and critical care environment and was developed to support rapid and immediate haemorrhage control in trauma patients but can also be used in patients with ruptured aneurysms of the abdominal aorta. Importantly, the ER-REBOA™ Catheter is indicated to be safely and effectively placed with or without the aid of medical imaging if none is available. The device will be placed via femoral artery directly in the thoracic part of the aorta, with the aid of a standard 7-F introducer sheath. For blood pressure monitoring standard equipment (transducer and 0.9% saline flush unit) are required.

Puncture of the femoral artery to gain access to the arterial system is a standard procedure in the emergency and critical care area, as well as in cardiology, interventional radiology, angiology/vessel surgery and anaesthesiology. Puncture itself can be difficult or impossible, even with the aid of ultrasonography, especially in an emergency. Nevertheless, even prehospital puncture of the femoral artery during cardiac arrest in order to obtain hemodynamic monitoring and guide CPR has shown feasible. Handling the balloon catheter requires a short introduction and some mannequin training before first use.

Preclinical Evidence Several studies have examined the effect of continuous balloon occlusion of the aorta during non-traumatic cardiac arrest in animal models. Occlusion of the aorta with and without selective aortic arch perfusion was shown to increases coronary artery blood flow and perfusion pressure as well as carotid perfusion pressure and blood flow, thus leading to improved rates of ROSC, 24h- and 48hsurvival and neurological function in animals. To the investigators' knowledge, no conflicting data failing to show the described effects has been published, leading to the suggestion that further research should concentrate on the question whether these promising findings apply for humans, too.

Clinical Evidence to Date Recent advances in technology have led to the endovascular approach to the aorta being no longer exclusively the domain of cardiology, angiology and vascular surgery, but emergency and critical care physicians and surgeons using the technique in the emergency and critical care setting as well as in a prehospital setting to control major pelvic and abdominal hemorrhage in trauma victims. Therefore, regarding the use of the ER-REBOA catheter, available literature reports mainly trauma victims, where endovascular occlusion of the aorta was used to control exsanguinating hemorrhage but was also shown to lead to meaningful increases of mean arterial blood pressure immediately following occlusion of the aorta. A recent study examining the outcome of trauma victims with severe hemorrhage also included patients in traumatic cardiac arrest and showed a neurological intact survival rate of 10%, whereas survival of cardiac arrest due to massive hemorrhage treated with emergency department thoracotomy with aortic cross-clamp is known to be dismal. Similarly, patients with non-traumatic hemorrhage mainly from intraabdominal aneurysmal rupture received REBOA until definitive hemorrhage control, with 7 of 11 patients being in cardiac arrest at the time of insertion and a high survival rate of 57%. Regarding cardiac arrest not associated with hemorrhage and/or trauma, for humans only case reports exist, describing neurological intact survival in one case of refractory cardiac arrest with PEA/Asystole during coronary angiography, where after 20 minutes of futile ALS an intra-aortal balloon pump (IABP) was inserted, with detection of ROSC 30seconds after occlusion of the descending aorta. Importantly, the estimated benefit of increased mean arterial pressure and coronary perfusion pressure even with intermittent occlusion of the aorta has led to the recommendation to use the IABP (after switching to a pressure-triggered mode) in patients with cardiac arrest after heart surgery and IABP in place.

Medical Device: Rationale for the intended purpose in study (pre-market MD) The ER-REBOA™ Catheter was chosen because it is (to the investigators' knowledge) the only REBOA catheter which can be inserted without a guide wire, and the placement does not necessarily need radiologic guidance.

Risks / Benefits As only patients will be included who have failed to respond to recommended standard resuscitation therapy (refractory cardiac arrest under BLS/ALS) and not qualifying for e-CPR, these patients can only gain the benefit of improved survival to hospital discharge and neurological good outcome, given the extremely poor chance of neurologic intact survival otherwise. This outweighs the risks associated with arterial puncture (damage to the vessel/ tissue, pseudoaneurysma, fistula, surgical repair after successful resuscitation) and the theoretical risk of limb paralysis after prolonged (> 2 hours) ischemia.

Survival of cardiac arrest with an unwanted unfavorable neurologic state is an inherent risk of resuscitation per se. Use of a REABOA device might possibly shift patients from the out-come groups "death" towards "vegetative state" or "home-bound and dependent on others". The investigators cannot estimate this specific "risk of survival", which, depending on personal beliefs, are not necessarily seen as bad outcome at all.

As described above, the ER-REBOA™ Catheter is intended for temporal occlusion of large vessels and specifically designed for the use in an emergency or intensive care setting, as it is planned in this study. Possible problems with malpositioning and injury to the access site, rarely requiring surgical repair, have been addressed. The extreme complication - the case of exsanguinating hemorrhage due to the puncture - is judged acceptable by the study group compared to the potential benefit of surviving otherwise refractory cardiac arrest during standard ALS.

Justification of choice of study population To evaluate the feasibility of the REBOA catheter placement during resuscitative efforts due to cardiac arrest, the investigators cannot perform the study in already deceased persons since the investigators need the hemodynamic measurements during CPR as a success parameter that measurable blood pressure can be generated in the aorta due to the occlusion. Since cardiac arrest and CPR cannot be performed in healthy subjects or in patients during routine cardiac surgery or coronary angiography, the investigators can only perform the study in patients suffering from actual cardiac arrest. Patients in cardiac arrest are per definition clinically dead (no circulation - no breathing) and in the most extreme life threatening emergency. Therefore patients in CA cannot consent beforehand. Standard CPR is a highly focused team-orientated and standardized event to save the life of the patient, and given the nature of cardiac arrest, an extremely time-sensitive emergency. It will therefore be no time to contact family members or next of kin to get consent for a study, and timely involvement of an independent physician in the study consent procedure beforehand will not be achievable in each case (despite the intend to do so). If the patient survives, a daily assessment of the patient's capacity to give informed consent will be done until the patient is discharged from the ICU, as in any case of significant clinical change. When the patient is judged capable of giving consent, a post hoc informed consent process will be performed as soon as possible. If the patient is permanently lacking capacity to consent and if no written statement of wishes formulated in a state of capacity is available, a proxy consent will be obtained from a person authorized to represent the patient as soon as possible, bearing in mind the emotional stress the proxy experienced after the event of sudden cardiac death and resuscitation and providing an appropriate time frame.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the resuscitation bay, intensive care unit or coronary angiography laboratory with refractory cardiac arrest, defined as failure to achieve stable ROSC within 10 min of fully established standard care (ALS), who do not qualify for extracorporeal cardiac life support (e-CPR).

Exclusion Criteria:

* Patients whose underlying disease limit survival and resuscitation measures are stopped after initial assessment, or evaluation reveals futile clinical situation

  * Patients with advanced directives or living will which excludes CPR
  * Age < 18 years (device certified >18 years)
  * Qualifying for other treatment options, namely eCPR (CPR with extracorporeal membrane oxygenation (ECMO) as life assist device)
  * Patients in whom no femoral arterial access site cannot accommodate a 7 Fr (minimum) introducer sheath
  * Known to have an aortic diameter larger than 32 mm
  * Evidence of thoracic hemorrhage (eFAST)
  * Study personnel and/or study equipment not available at the time of study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Percentage of successful placements | 10 minutes
  Percentage of successful placements within 10 minutes from start of the investigated procedure (start defined as end of skin disinfection) to balloon inflation

SECONDARY OUTCOMES:
Number of attempts | 60 min
  Number of attempts (both vessel puncture and placement of catheter),
Time of the successful attempt | 60 min
  Time of the successful attempt (from successful arterial puncture to balloon inflation),
Overall time | 60 min
  Overall time (from start to inflation)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Levis, MD, Principal Investigator — Dep of Intensive Care Medicine, University Hospital Bern
Locations (1):
- Departement of Intensive Care Medicine - University Hospital Bern - Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
individual decision upon request